CLINICAL TRIAL: NCT01398150
Title: Cranberry Enhances Human Immune Function and Reduces Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Ocean Spray, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CB-79545
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2010-02

CONDITIONS: Healthy Humans
Keywords: gamma delta T cell; proliferation; cytokine secretion; immune function; antioxidant status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sweetened Beverage (Placebo Comparator): looks like and is given in the same way as the experimental treatment but contains no active ingredient
  Interventions: Dietary Supplement: Beverage made to look like the cranberry beverage
- Cranberry Beverage (Experimental): 15 ounce bottle of cranberry beverage consumed daily for 70 days
  Interventions: Dietary Supplement: Beverage made from cranberry compounds

INTERVENTIONS:
Dietary Supplement: Beverage made to look like the cranberry beverage — one 15 ounce bottle of beverage consumed daily
  Arms: Sweetened Beverage
Dietary Supplement: Beverage made from cranberry compounds — one 15 ounce bottle consumed daily for 70 days
  Arms: Cranberry Beverage

SUMMARY:
The purpose of this study is to determine whether consuming a beverage made with cranberry polyphenols and proanthocyanidins is effective in modifying immune function by enhancing immune cell proliferation, cytokine production, and antioxidant capacity. If immune cell proliferation is improved, the subjects are expected to have fewer cold and flu symptoms.

DETAILED DESCRIPTION:
The study will be conducted as a randomized, double blind, placebo-controlled parallel trial. Subjects will be randomly assigned to either the Treatment (cranberry beverage) group or the Placebo group and each will be instructed to consume the test beverages twice a day for 70 days. The beverage is not commercially prepared juice, but is a beverage prepared with an extract of cranberry that contains polyphenols and proanthocyanidins. Blood is taken at baseline, and day 70. Subjects are given a diary to keep a record of their cold and flu symptoms. Serum is used to determine the antioxidant activity by the ORAC method. Peripheral blood mononuclear cells are isolated from the blood draw and used fresh, cultured for 24 hours or cultured for 10 days. Freshly isolated cells will be used to determine αβ-T, γδ-T, B and NK cell numbers and then cultured in autologous serum for 10 days to determine how well they proliferate. The supernatant of 24 hour cultures will be used for cytokine determination. If cells have been primed by the beverage made with cranberry compounds, the investigators expect the cells to proliferate to a greater extent and have modified cytokine production compared to placebo. If the beverage made with cranberry compounds enhances the proliferation of one or more of these cell types (αβ-T, γδ T, B or NK cell), then it is possible that there will be fewer cold and flu symptoms in the group consuming the cranberry beverage. Incidence of illness is not expected to change, only the severity of the illness.

ELIGIBILITY:
Inclusion Criteria:

* Health male or non-pregnant female
* Between the ages of 21 and 50
* BMI between 18 and 35

Exclusion Criteria:

* High blood pressure define as 140/90
* Ongoing or chronic illness or infection
* On hypertensive medication, immunosuppressive drugs, antibiotics, or chronic use of NSAIDS
* Taking plant-based dietary supplements, antioxidant supplements, or probiotics
* Vegetarian or strict vegan
* Consume more than 1 cup of tea (iced or hot) per day
* Consumes more than 2 glasses of alcoholic beverages per day
* Consume more than 7 fruits and vegetables per day

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Physiological modifications to immune cell function | 70 days
  Proliferation of γδ-T cells when cultured ex vivo in autologous serum

SECONDARY OUTCOMES:
Cold and flu symptoms | 70 days
  Incidence and severity of cold and flu symptoms, total and individual. Other signs of severity, for example, visits to doctor or health clinic, reduction in daily activities, medications prescribed or purchased OTC.
Anti-inflammatory outcome | 70 days
  Serum antioxidant status, cytokine production and proliferation of αβ-T, B and NK cells

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Percival, PhD, Principal Investigator — University of Florida
Locations (1):
- 449 Food Science and Human Nutrition Department, Gainesville, Florida, United States

REFERENCES:
- [Derived] Nantz MP, Rowe CA, Muller C, Creasy R, Colee J, Khoo C, Percival SS. Consumption of cranberry polyphenols enhances human gammadelta-T cell proliferation and reduces the number of symptoms associated with colds and influenza: a randomized, placebo-controlled intervention study. Nutr J. 2013 Dec 13;12:161. doi: 10.1186/1475-2891-12-161. PMID 24330619